CLINICAL TRIAL: NCT05585710
Title: Pulsed Lavage in Implant-Based Breast Reconstruction: A Randomized Control Trial
Brief Title: Pulsed Lavage in Implant-Based Breast Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Richard Jobe Fix, Professor in the Department of Plastic Surgery, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300009900
Record Dates: First submitted 2022-10-14; First posted 2022-10-19 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Breast Reconstruction
Keywords: breast reconstruction; implant-based breast reconstruction; pulsed lavage
MeSH Terms: interventions — Mastectomy, Simple; Tissue Expansion Devices

STUDY DESIGN:
Intervention Model Description: Two cohorts will be established. One cohort will include patients who undergo pulsed lavage to wash out the mastectomy pocket. The other cohort will include patients who do not receive pulsed lavage.
Masking Description: Pulsed Lavage is a surgical technique that cannot be masked from the investigators performing the operation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pulsed Lavage Washout (Experimental): This cohort will undergo standard of care bilateral or unilateral mastectomies as determined by breast surgical oncologists and immediate standard of care breast reconstruction with tissue expander placement and pulsed lavage washout.
  Interventions: Other: Pulsed Lavage Washout; Procedure: Implant-based breast reconstruction; Procedure: Bilateral or unilateral mastectomy; Device: Tissue expander; Other: Acellular dermal matrix
- No Pulsed Lavage (Active Comparator): This cohort will undergo standard of care bilateral or unilateral mastectomies as determined by breast surgical oncologists and immediate standard of care breast reconstruction with tissue expander placement.
  Interventions: Procedure: Implant-based breast reconstruction; Procedure: Bilateral or unilateral mastectomy; Device: Tissue expander; Other: Acellular dermal matrix

INTERVENTIONS:
Other: Pulsed Lavage Washout — Use of pressurized, pulsed triple antibiotic solution to irrigate mastectomy pocket
  Arms: Pulsed Lavage Washout
Procedure: Implant-based breast reconstruction — Standard of care; use of triple antibiotic solution delivered via bulb syringes to irrigate mastectomy pocket
Procedure: Bilateral or unilateral mastectomy — Standard of care
Device: Tissue expander — Standard of care
Other: Acellular dermal matrix — Standard of care

SUMMARY:
To determine if there is any benefit to using pulsed lavage to wash out the mastectomy pocket during breast reconstruction. Primary outcomes will include post-op complications including surgical site infection (SSI), hematoma, seroma, and implant failure.

DETAILED DESCRIPTION:
After being informed of the study including potential risks and benefits, all patients giving consent who meet eligibility requirements will undergo randomization into either the pulsed lavage arm (receive mastectomy pocket wash out using pulsed lavage) or the no pulsed lavage arm (pulsed lavage will not be used). Randomization will occur using a random number generator with even numbers resulting in a pulsed lavage washout and odd numbers resulting in no pulsed lavage washout.

The patients will be followed in clinic for a maximum of 3 months to evaluate the surgical site. The two cohorts will be compared at the end of the study to determine whether there is any benefit to using pulsed lavage to wash out the mastectomy pocket during breast reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Between 18 and 75 years of age, inclusive
* Undergoing implant-based breast reconstruction (unilateral or bilateral) with immediate expander at mastectomy
* Able to understand and willing to sign an Institutional Review Board (IRB) approved written informed consent document

Exclusion Criteria:

* Male
* < 18 years of age or > 75 years of age
* Undergoing implant-based breast reconstruction (unilateral or bilateral) with delayed expander at mastectomy

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Post-op Complications | up to 3 months
  unintended complications that occur post-surgically

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Fix, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No